CLINICAL TRIAL: NCT07404774
Title: Prospective Evaluation of Hemorrhoid Suture Mucopexy (SM) Combined With Laser Hemorrhoidoplasty (LHP) for Symptomatic Hemorrhoidal Disease: A Cohort Study
Brief Title: Hemorrhoid Suture Mucopexy Combined With Laser Hemorrhoidoplasty
Acronym: HeMuLa
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, George Theodoropoulos, Professor, National and Kapodistrian University of Athens
Other Study IDs: 100/22-12-2025
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Haemorrhoid; Haemorrhoidal Bleeding; Anorectal Surgeries; Anorectal Diseases
Keywords: haemorrhoid; laser; mucopexy; suture mucopexy; LHP; haemorrhoidoplasty
MeSH Terms: conditions — Hemorrhoids; Rectal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laser Haemorrhoidoplasty and Suture Mucopexy — The procedure combines laser ablation (LHP) with suture mucopexy (SM) performed without Doppler guidance.
  Suture Mucopexy (SM): Using a slotted proctoscope, continuous suture mucopexy (plication) is performed at standardized anatomical positions (typically 4, 7, 11 o'clock) to lift the prolapse and ligate feeding vessels. Sutures are placed approximately 2-4 cm proximal to the dentate line.
  Laser Hemorrhoidoplasty (LHP): A 1470nm diode laser fiber is inserted into the hemorrhoidal cushion. Energy is delivered (approx. 250-350 J per pile) to induce shrinkage and fibrosis.

SUMMARY:
This prospective cohort study evaluates whether combining "suture mucopexy" (a simple stitch-based lift of prolapsed tissue) with Laser Hemorrhoidoplasty (LHP) can effectively relieve pain, bleeding and prolapse in adults with moderate-to-severe hemorrhoids (Grades II-IV). Participants will undergo the combined, non-Doppler-guided procedure and be followed for one year. The primary question is how long patients need post-operative pain medication and if they first experience complete symptom relief; secondary questions examine quality-of-life, safety (bleeding, urinary retention, stenosis) and the rate of hemorrhoid recurrence/re-operation.

DETAILED DESCRIPTION:
Laser Hemorrhoidoplasty (LHP) offers a minimally invasive option for symptomatic hemorrhoids, yet in advanced disease (Goligher III/IV) recurrence rates of 20-35 % have been reported because residual mucosal prolapse persists. Adding a suture-based mucopexy (SM) eliminates the prolapse and ligates feeding vessels without the need for Doppler guidance, thereby potentially reducing recurrence while preserving the low-pain advantage of LHP. Preliminary experience with 50 patients at this centre demonstrated feasibility, low early complication rates, and promising symptom control, justifying a formal prospective evaluation.

The present study is a single-center, prospective observational cohort enrolling consecutive eligible adults over a 24-month accrual period. All participants receive the same combined LHP + SM technique; no comparator arm is planned. Follow-up visits occur at postoperative week 6, month 6 and month 12.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years).
* Symptomatic Hemorrhoidal Disease (Goligher Grades II, III, IV).
* Patients with or without recurrent disease after prior procedures (e.g., RBL, infrared coagulation, Milligan-Morgan, etc).

Exclusion Criteria:

* Acutely thrombosed hemorrhoids.
* Concomitant anal fistula or abscess requiring separate surgical management.
* IBD (Crohn's/Ulcerative Colitis) with active rectal involvement.
* Previous Stapled Haemorrhoidopexy (SH/Longo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be drawn from the outpatient and surgical patient base of the Department of Colorectal Surgery at Ippokrateio University Hospital. All individuals presenting with symptomatic hemorrhoidal disease of Goligher Grades II-IV, regardless of prior non-excisional treatment, are eligible for invitation to the study. This cohort represents a real-world clinical population of patients undergoing minimally invasive hemorrhoid management within a single, high-volume colorectal surgery practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | perioperatively
  Defined as the number of days from surgery until the complete cessation of all opioid and non-opioid pain medications.
Primary Symptom Relief | perioperatively
  Patient-reported cessation of bleeding and/or pain.

SECONDARY OUTCOMES:
Nyström Hemorrhoid Severity Score (HSS) | 12 months
  5 items (pain, itching, bleeding, prolapse, soiling) scored 0-3 (higher score indicates worse symptoms), assessed at preoperative baseline, 6 weeks, 6 months, and 12 months.
Morbidity | 3 months
  Postoperative morbidity (Clavien-Dindo classification), ranging from Grade I (minor, no intervention) to Grade V (death), at 30 days and 90 days.
Complications | 12 months
  Postoperative complications, specifically tracking urinary retention, bleeding, and anal stenosis (yes/no)
Reoperation Rate | 12 months
  Need for secondary surgical intervention for recurrence or complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Ippokrateio Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided